CLINICAL TRIAL: NCT01111695
Title: Open Label Study (Phase 2) to Evaluate the Safety, Tolerance and Efficacy of a Ionic Silver and Honey Preparation to Treat Chronic Wounds of the Lower Legs
Brief Title: Evaluation of a Ionic Silver and Honey Preparation to Treat Chronic Wounds of the Lower Legs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Haute école de santé - Genève (Unknown)
Responsible Party: Dr Denis SALOMON/ Médecin adjoint agrégé, Service de dermatologie - HUG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER 09-013
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-02

CONDITIONS: Leg Ulcer
Keywords: wound healing; granulation tissue; Varicose Ulcer
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Honey and ionic silver dressing (Experimental)
  Interventions: Device: ApisSept

INTERVENTIONS:
Device: ApisSept — honey and ionic silver based dressing

SUMMARY:
In this open study, the primary objective is to study the efficacy and clinical outcome of the chronic wounds treated with this preparation for 8 weeks on 30 adults. Evaluation will be based on standardised photographs and clinical data.

The secondary objectives are to evaluate the tolerance and side effects of the honey based preparation in the management of chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Chronic wounds due to arterial or venous insufficiency stages 1 to 3 and difficult to heal with the usual treatments and
* Written informed consent

Exclusion Criteria:

* Refuse to give written informed consent.
* Patient suffering from mental disorder that may interfere with the treatment.
* Known allergy or intolerance to any of the products used in the formulation.
* Having received systemic antibiotics within 7 days of starting treatment with honey based formulation.
* Arterial insufficiency stage IV of the lower limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Granulation and /or epithelial tissue progression | 8 weeks
  Granulation and /or epithelial tissue progression as observed by standardised photography (colour-based and analysis of the wound).

SECONDARY OUTCOMES:
Tolerance | 8 weeks
  Tolerance: Evaluate for signs and symptoms of irritation,inflammation, allergy or pain in and around the treated zone by clinical observation.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Salomon, Dr, Principal Investigator — University Hospital, Geneva
Locations (1):
- Home Care Service of the canton of Geneva, Geneva, Switzerland